CLINICAL TRIAL: NCT04094831
Title: Community-based Screening to Determine the Prevalence, Current Health and Nutritional Status of Individuals With Chronic Kidney Disease (CKD) and Measure the Outcome of Health Education to Enhance Knowledge, Awareness and Risk Reduction Strategies in Mirzapur Sub-district, Bangladesh
Brief Title: Community-based Screening of Chronic Kidney Disease (CKD) and Measure the Impact of Health Education
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Hiroshima University (Other); Child Health Research Foundation, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: PR-19081
Record Dates: First submitted 2019-09-17; First posted 2019-09-19 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-01

CONDITIONS: Chronic Kidney Disease (CKD)
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Active Comparator): Intervention group (Health education through CKD campaign and mHealth) technology
  Interventions: Other: Health education
- Control (Active Comparator): No intervention
  Interventions: Other: Health education

INTERVENTIONS:
Other: Health education — The intervention group will receive health education through CKD campaign and mHealth technology. During the half day CKD campaign, health education materials (leaflet and short textbook and recording notebook) will be provided to the study participants. A nephrologist will facilitate the campaign and contents (Annex-3) of the text book and leaflet (Annex-4) will be discussed. Important message from the text book (such as stage, risk factor, preventive measures) will be used to develop the leaflet. In addition,Basic health education information about CKD is included in the contents to help patients gain knowledge, awareness, and improve their behaviors. Discussion on basic kidney diseases, risk factors, and preventive measures of CKD is performing by CHWs over a mobile phone call to the study patients. The patients have the liberty to discuss their health-related issues with the CHWs over a period of 10 minutes

SUMMARY:
Background: Chronic kidney disease (CKD) is a global public health concern. Currently 10-16% adults are affected with CKD. Adult individuals from low- and middle-income countries are at higher risk of developing CKD and End stage renal disease (ESRD). Preventive and risk reduction measures have potentials to reduce the disease progression; however, population in general from developing countries are yet to be properly aware about all these strategies that may help reduction in progression of CKD.

Knowledge gap: Specific studies are grossly lacking about CKD prevalence, its associated factors, and the knowledge and awareness about preventive and risk reduction strategies among adults with CKD in rural and peri-urban Bangladesh. Moreover, knowledge gaps still exist about the role of Protein Energy Wasting (PEW), physical activities, medication adherence, dietary practice, salt restriction behaviours, etc. in influencing progression of CKD.

Relevance: It has become essential to know more about the burden of CKD, its associated factors, current knowledge and awareness about healthy practices related to CKD and formulation of appropriate preventive and risk reduction strategies that will have potentials in reducing the progression of CKD in rural and peri-urban Bangladesh. The health education program for population in general and CKD individuals in particular will help in achieving meaningful results.

Hypothesis:Health education about CKD and its preventive and risk reduction strategies will enhance the knowledge, awareness, and motivation for healthy practices among the residents of demographic surveillance system (DSS) area with CKD.

Objectives:

To implement and evaluate impact of a health education program in order to enhance knowledge, awareness, and motivation about healthy practices among rural adults suffering from CKD.

Methods:

A community based randomized controlled effectiveness trial (RCT) Study site: DSS area of Mirzapur sub-district under Tangail, Bangladesh.

Outcome measures:

Primary outcomes: Changes of scores of Australian CKD knowledge questionnaire Secondary outcomes: Awareness, Quality of life (QOL), and healthy practices leading to maintenance of blood pressure, blood sugar and body weight within normal ranges by the adult CKD individuals.

DETAILED DESCRIPTION:
This would be a community-based randomized controlled trial (RCT) among the individuals diagnosed as having CKD with stage 1-3 who agreed to participate.

Registration/Enrolment of participants:

Community health workers (CHWs) will perform home -visits to obtain written informed consent, perform physical examination, and interview the respondents administering field tested questionnaires.

Interviewing by administering a structured questionnaire: if changed from Study 1: Age, gender, marital status, occupation, educational background, income/month, participant's current medical history including medication use, past medical history, sleeping hours, and family history (3rd generation) including current and immediate past medical history.

Physical examinations will be performed to measure: Blood pressure, pulse, height, weight, waist circumference, hip circumference, triceps skin fold (TSF), mid-upper arm circumference (MUAC), body mass index (BMI) and mid-arm muscle circumference (MAMC).

Blood sample (at hospital) Serum creatinine (estimate eGFR), serum albumin, Hb%, FBS, HbA1C, lipid profile (TP, HDL-c, LDL-c, triglyceride, and ratio: estimate non-HDL), serum uric acid, Urea (BUN).

Urine specimens (at hospital) Albumin to creatinine ratio (ACR), urine RME, urine Na (calculate sodium intake)

Questionnaires/Interviewing :

Chronic Kidney Disease Knowledge Questionnaire (24 questions) Awareness question (1 question) QOL (5 EURO-QOL questionnaire) Randomisation: A simple randomization (1:1) either intervention group or control group will be undertaken following a computer-generated random number sequence. An experienced statistician, who will not be involved in the study in any way, will prepare the randomization table and list of study participants' numbers with corresponding intervention allocations for CKD individual in serially numbered sealed envelopes according to randomization schedule to correspond to the serial number of the CKD individuals. These envelopes will be kept in an office locker. Allocation will be concealed in identical sealed envelopes that will only be opened when the study participant is ready for enrolment. This will take place after a CKD individual has been enrolled in the study following obtaining voluntarily informed written consent and assigning a study number. Necessary attempts will be made to keep CHWs unaware about case/control status of the participants. Similar approach will also be followed at the time of data analysis.

Study contents:

The intervention group will receive health education through CKD campaign and mHealth technology. During the half day CKD campaign, health education materials (leaflet and short textbook and recording notebook) will be provided to the study participants. A nephrologist will facilitate the campaign and contents (Annex-3) of the text book and leaflet (Annex-4) will be discussed. Important message from the text book (such as stage, risk factor, preventive measures) will be used to develop the leaflet. In addition, education through mHealth will be provided by Short Message Service (SMS) during the study period. The contents of the SMS are: 1). Reduce salt intake; 2) Do exercise and take medicine regularly; 3). Control blood pressure (if hypertensive) and blood sugar (if diabetic); and 4) Avoid painkiller and smoking will be sent to the participants using mobile phone once a week for first 2.5 months and once a 2-week for next 3 months.

The CKD knowledge questionnaire consisted a total of 24 questions with the multiple-choice options 'true', 'false' and 'I don't know'. The validated questionnaire will be adapted according to Bangldesh context and will be pre-tested before starting the study. The quality of life will be assessed using an adapted and validated Bangla version of the 5 EURO-QOL questionnaire. It has five domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.

Sample size calculation:

Assuming that proportion of knowledge and awareness among CKD patients at baseline as 30%; and at the end of six months it will increase to 70% (intervention group) and 40% (control group). Therefore, considering 90% power and 20% loss to follow-up the total sample size will be 136 (68 in each group).

Data analysis:

The descriptive statistics will be expressed as frequency, mean, median, cross tabulation, and standard deviation. Chi-square test, t-test or Mann-Whitney U-test will be performed to see the differences between intervention group and control group at baseline, 3 and 6 months. Multiple comparisons will be performed by ANOVA test for evaluation of the outcome variables such as CKD knowledge and awareness questionnaire and QOL at baseline, 3 and 6 months. Data will be analyzed using SPSS ver. 22.0 (IBM Co., Armonk, NY) and the significance level will be set at the level of p < 5%.

ELIGIBILITY:
Inclusion Criteria:

1. All diagnosed CKD patients with stage 1-3 from Study 1
2. Who gave written informed consent to participate in the study.
3. At least 1-5 years of schooling
4. Using mobile phone at house

Exclusion Criteria:

1. CKD participants with stage 4-5.
2. Not willing to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Chronic Kidney Disease Knowledge Questionnaire | 6 months after the intervention
  The questionnaire consisted a total of 24 questions with the multiple-choice options 'True', 'False' and 'I don't know'. Correct responses were given a score of 1 and incorrect responses were given a score of 0. The option 'I don't know' was considered as lack of knowledge and given a score of 0.
  Score <50% considered as poor. The questionnaire consisted a total of 24 questions with the multiple-choice options 'True', 'False' and 'I don't know'. Correct responses were given a score of 1 and incorrect responses were given a score of 0. The option 'I don't know' was considered as lack of knowledge and given a score of 0.
  Score <50% considered as poor.

SECONDARY OUTCOMES:
EURO- Quality of Life questionnaire (5 EURO-QOL questionnaire) | at 3 months and 6 months of intervention
  This questionnaire based on 5 Dimensions, five-level version questionnaire. This scale is numbered from 0 to 100. 100 mean the best health you can imagine.

CONTACTS AND LOCATIONS:
Locations (1):
- icddr,b Mirzapur Field site, Tāngāil, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sarker MHR, Moriyama M, Rashid HU, Rahman MM, Chisti MJ, Das SK, Saha SK, Arifeen SE, Ahmed T, Faruque ASG. Chronic Kidney Disease Awareness Campaign and Mobile Health Education to Improve Knowledge, Quality of Life, and Motivation for a Healthy Lifestyle Among Patients With Chronic Kidney Disease in Bangladesh: Randomized Controlled Trial. J Med Internet Res. 2022 Aug 11;24(8):e37314. doi: 10.2196/37314. PMID 35969429
- [Derived] Sarker MHR, Moriyama M, Rashid HU, Rahman MM, Chisti MJ, Das SK, Jahan Y, Saha SK, Arifeen SE, Ahmed T, Faruque ASG. Health Education Through a Campaign and mHealth to Enhance Knowledge and Quality of Life Among Patients With Chronic Kidney Disease in Bangladesh: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2021 Nov 19;10(11):e30191. doi: 10.2196/30191. PMID 34806998